CLINICAL TRIAL: NCT00648895
Title: Effect of Nebivolol on Forearm Vasodilation, Nitric Oxide Bioavailability, and Oxidative Stress in Patients With Stage 1/2 Hypertension
Brief Title: A Study of the Effect of Nebivolol to Evaluate Its Vasodilatory Effects in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: John Whalen, MD, Executive Director, Clinical Development, Cardiovascular, Forest Research Institute, a subsidiary of Forest Laboratories Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB-MD-08
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Results first posted 2010-09-20 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-08

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure; Nebivolol; Bystolic (TM); Metoprolol ER (TM)
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Nebivolol
  Interventions: Drug: Nebivolol
- 2 (Active Comparator): Metoprolol ER (TM)
  Interventions: Drug: Metoprolol ER (TM)

INTERVENTIONS:
Drug: Nebivolol — nebivolol 10mg, 20mg, 40mg daily dosage, oral administration
  Other Names: Bystolic (TM)
  Arms: 1
Drug: Metoprolol ER (TM) — Metoprolol ER 100mg, 200mg, 400mg, daily dosage, oral administration
  Other Names: Toprol XL (TM)
  Arms: 2

SUMMARY:
The study is designed to compare the effects of nebivolol (10, 20, 40mg/day) with another beta blocker, extended-release metoprolol, at a range of doses. Its purpose is to study the mechanism of action of nebivolol on forearm blood flow, nitric oxide availability and other biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ambulatory outpatients 18-79 years old at screening
* Minimum 2-year history of Stage I/II hypertension
* Qualifying blood pressure criteria for study entry and for randomization
* Willing to adhere to the dietary compliance and undergo protocol procedures
* Have a lifestyle that will permit him/her to attend all evaluations, including those conducted on consecutive days

Exclusion Criteria:

* Have any form of secondary hypertension
* Have clinically significant respiratory or cardiovascular disease
* Presence/history of coronary artery disease or peripheral vascular disease
* Have diabetes mellitus, Type I or II
* Have a history of hypersensitivity to nebivolol, metoprolol, or any beta-blocker

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Lukic, MD., M.Sc., Study Director — Forest Research Institute, Inc., a Subsidiary of Forest Laboratories, Inc.
Locations (1):
- Forest Investigative Site, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from November 2007 to May 2009 at one US location.
Pre-assignment Details: All patients went through a 4-5 week, single blind, placebo washout phase before randomization.
Groups:
- Nebivolol: A 6-week up-titration period (the dose of nebivolol was increased from 10 mg/d to a maximum of 40mg/d, if necessary, to achieve hypertension control) followed by a 4-week stable-dose period and a 2-week down-titration phase
- Metoprolol ER (TM): A 6-week up-titration period (the dose of metoprolol ER was increased from 100 mg/d to a maximum of 400mg/d, if necessary, to achieve hypertension control) followed by a 4-week stable-dose period and a 2-week down-titration phase.
Period: Overall Study
Arm/Group | Nebivolol | Metoprolol ER (TM)
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Metoprolol ER (TM) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 2 | 5 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 59.5 (5.8) | 67.3 (11.6) | 63.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline to End of Treatment for the Difference Between the Post-ischemia and Pre-ischemia Forearm Vascular Resistance (FVR).
Description: Pre-and post-ischemia forearm vascular resistance (FVR), calculated by forearm blood flow (FBF) and systolic blood pressure (SBP), and assessed at the trough/pre-meal time point (used for percentage change analysis between baseline and postbaseline). Measurements occured at baseline (visit 5) and end of treatment (week 10).
Time Frame: Before treatment and after 10 weeks
Population: Due to the small sample size, no efficacy conclusion could be made. 0 measured value primary outcome =Not applicable.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Nebivolol | Metoprolol ER (TM)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 months
Arm/Group | Nebivolol | Metoprolol ER (TM)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=6) | Metoprolol ER (TM) (N=6)
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early because of difficulties with enrollment. Only 12 of 30 planned patients were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & can embargo communications re: results for 60 days from time submitted to sponsor for review. PI shall not disclose sponsor's confidential information. Upon sponsor's request, PI shall delete any proprietary info & shall not include raw data in the publication. On sponsor's request, PI shall delay submission for any pub while sponsor files patent applications. Any publication will give recognition to Sponsor's support.